CLINICAL TRIAL: NCT01430026
Title: Efficacy and Complication of Gentamicin Nasal Irrigation in Chronic Rhinosinusitis
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: 004/2554(EC3)
Record Dates: First submitted 2011-09-05; First posted 2011-09-07 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Sinusitis
Keywords: chronic sinusitis; gentamicin nasal irrigation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The propose of this study to determine efficacy and complication of gentamicin nasal irrigation in chronic rhinosinusitis

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is characterized by symptoms > 12 weeks

Two or more symptoms one of which should be either nasal blockage /obstruction/congestion or nasal discharge (anterior/posterior nasal drip):

* facial pain/pressure
* reduction or loss of smell)

Mainstay of treatment are medical and surgical treatment ( ATB, adenoidectomy, ESS) Adjunctive treatment : normal saline nasal irrigation, nasal corticosteroids, nasal decongestants, mucolytics Topical antibiotic therapy in patients with refractory sinusitis has been shown to improve symptoms, quality of life, and mucosal aspect Nasal lavage with Mupirocin represent an effective and well tolerated alternative treatment of surgically recalcitrant chronic rhinosinusitis

In pediatrics allergy clinic at Siriraj hospital since 2006 use Gentamicin nasal irrigation for chronic rhinosinusitis.There have been no studies in gentamicin irrigation in chronic rhinosinusitis. The aims of this study are to evaluate:

1. Efficacy of gentamicin nasal irrigation in chronic rhinosinusitis (outcomes: frequency of sinusitis, frequency of antibiotic usage)
2. Complication of gentamicin nasal irrigation usage

ELIGIBILITY:
Inclusion Criteria:

* Chronic rhinosinusitis patients who were followed in pediatrics allergy clinic at Siriraj hospital between January 1, 2005, and February 28, 2011
* Gentamicin nasal irrigation usage for longer than 3 months

Exclusion Criteria:

* Patients who used azithromycin prophylaxis within 1 year before and 6 months after started gentamicin nasal irrigation
* Patients received IVIG within 1 year before and 6 months after started gentamicin nasal irrigation
* Patients underwent endoscopic sinus surgery within 1 year before and 6 months after started gentamicin nasal irrigation
* Patients received IT within 1 year before and 6 months after started gentamicin nasal irrigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric allergy clinic in siriraj hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Frequency of sinusitis | 1 year

SECONDARY OUTCOMES:
Complications of gentamicin nasal irrigation usage | 1 year
Frequency of antibiotic usage | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nualanong Visitsunthorn, professor, Principal Investigator — Department of Pediatrics Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Fokkens W, Lund V, Mullol J; European Position Paper on Rhinosinusitis and Nasal Polyps group. European position paper on rhinosinusitis and nasal polyps 2007. Rhinol Suppl. 2007;20:1-136. PMID 17844873
- [Background] Desrosiers MY, Salas-Prato M. Treatment of chronic rhinosinusitis refractory to other treatments with topical antibiotic therapy delivered by means of a large-particle nebulizer: results of a controlled trial. Otolaryngol Head Neck Surg. 2001 Sep;125(3):265-9. doi: 10.1067/mhn.2001.117410. PMID 11555764
- [Background] Uren B, Psaltis A, Wormald PJ. Nasal lavage with mupirocin for the treatment of surgically recalcitrant chronic rhinosinusitis. Laryngoscope. 2008 Sep;118(9):1677-80. doi: 10.1097/MLG.0b013e31817aec47. PMID 18545212